CLINICAL TRIAL: NCT04712240
Title: A Single Center Study Validating Accuracy of a Continuous Respiratory Rate Measurement Derived From a Respiratory Rate Monitoring Device (RRM): A Comparison With Capnography
Brief Title: Validating the Accuracy of a Continuous Respiratory Rate Measurement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REB20-2237
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Validation of Respiratory Rate Monitor Versus Capnography
Keywords: Respiration rate; Capnography; Continuous respiration rate monitoring

STUDY DESIGN:
Intervention Model Description: Participants will wear a portable respiration rate monitor that records respiration rate continuously while their respiration rate is also concurrently monitored and recorded using capnography (gold standard)
Masking Description: Participant, care giver, investigator and outcomes assessor will be aware that all participants are wearing a portable respiration rate monitor whose measurements will be compared to the gold standard of capnography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiration rate monitor (concurrently measured with standard of care capnography) (Other): Single group study whereupon participants will be fitted with portable respiration rate monitor around their chest for duration of surgery. Respiration rates acquired by the respiration rate monitor will be compared to capnography, which is standard of care and applied to all surgical cases
  Interventions: Device: Respiration rate monitor

INTERVENTIONS:
Device: Respiration rate monitor — A portable continuously monitoring respiration rate monitor will be fitted to each participant. The respiration rate monitor is housed within a comfortable chest strap that be secured to the participant for the duration of the surgical procedure

SUMMARY:
While respiratory rate is considered a critical vital sign, it often goes unmeasured or is ignored primarily due to shortcomings of the currently used measurement methods. Respiratory rate provides important information on a person's health condition and physiological stability, and an abnormal respiratory rate is a strong indicator that a health crisis is imminent. In fact, a sudden change in respiratory rate is one of the strongest predictors of mortality. Current techniques of monitoring respiratory rate have drawbacks that limit the frequency and convenience of the respiratory monitoring. Recognizing that closer respiration monitoring can save lives and improve quality of life, reduce hospital stays, and lower medical costs, the health care industry is seeking improved respiration monitoring products. The allocation of high-risk patients to intensive care for more careful monitoring or after surgery is often arbitrary, and such care might not be available routinely. For those patients who are cared for in 'general' wards where staffing levels are limited, a practical continuous monitor of respiratory rate would be of great value. This study will act as a pilot to determine the feasibility of using respiratory sensor device to monitor respiratory rate in hospitalized patients.

Deriving a measurement of respiratory rate from a respiratory rate monitoring (RRM) device is a technological approach that may overcome these limitations. The device principle is based on a piezoelectric sensor where chest expansions and contractions generate very small amounts of current by the piezoelectric sensor. The expansion and contractions are measured very accurately by over-sampling, filtering and digital signal processing to remove noise and any bias generated by the piezoelectric sensor itself or the sampling circuitry.

The study will be conducted from March 2021 to September 2021. During the first phase a convenience sample of 30 patients undergoing general anesthesia with muscle paralysis and mechanical ventilation will be recruited. This phase will help to validate the RRM against capnography in mechanically ventilated patients with a set respiratory rate. Following the first phase, 120 patients undergoing a procedure using sedation or spinal anesthesia will be recruited. Patients will be breathing spontaneously, and the respiratory rate will be monitored by capnography connected to the face mask or nasal prongs. Respiratory rate detected by capnography is recorded in the electronic medical records on a minute to minute interval.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants >= 18 years of age scheduled for elective surgery
* American Society of Anesthesiologists' Status Score <=3

Exclusion Criteria:

* Patients undergoing emergency surgery
* Patients undergoing abdominal procedures requiring skin prep of the lower chest area
* Patients undergoing breast surgery
* Patients undergoing shoulder surgery
* Patients with skin irritation in the area of monitor application
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Percentage of paired respiration rates within one breath per minute | Respiration will be measured during the duration of participants' surgical procedure
  Percentage of respiration rates measured by respiratory rate monitor that are within one breath per minute as measured by capnography

SECONDARY OUTCOMES:
Mean bias of errors | Respiration will be measured during the duration of participants' surgical procedure
  Mean bias of errors between respiration rates measured with respiratory rate monitor versus capnography
Standard deviation of errors | Respiration will be measured during the duration of participants' surgical procedure
  Standard deviation of errors between respiration rates measured with respiratory rate monitor versus capnography
Root mean square deviation of respiratory rate measurements | Respiration will be measured during the duration of participants' surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- South Health Campus, Calgary, Alberta, Canada